CLINICAL TRIAL: NCT01404286
Title: The Effects of a Session of Resistance Training on Sleep Patterns in the Elderly
Brief Title: Resistance Training and Sleep in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Centro de Estudos em Psicobiologia e Exercício (Unknown); Centro de Estudo Multidisciplinar em Sonolência e Acidentes - CEMSA (Unknown); Instituto do Sono (Unknown); Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Marco Tulio de Mello, Universidade Federal de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1059/06
Record Dates: First submitted 2011-05-24; First posted 2011-07-28 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2008-01

CONDITIONS: SLEEP DISTURBANCES Nec in ICD9CM
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- physical exercise (Experimental): Experimental group: physical exercise Control group: no physical exercise
  Interventions: Behavioral: Physical exercise
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Physical exercise — After the adaptation sessions, volunteers underwent a session of resistance training at 60% of 1 RM organized as follows: 3 sets of 10 to 12 repetitions on each exercise machine with a 1 minute and 30 second interval between each set and an interval of 2 minutes between each exercise machine, giving a total duration of training between 50 and 60 minutes. The sequence of exercise machines used was alternated by body segment. The sessions were performed at the same time of day (morning) under controlled temperature conditions (24 ± 21C).
  Other Names: Resistance Training; Sleep Patterns
  Arms: physical exercise

SUMMARY:
Purpose: The objective of this study was to evaluate the influence of a session of resistance training on the sleep patterns of elderly people.

Methods: Forty men aged 65 to 80 years, sedentary and clinically healthy were divided into two groups: the control group (n=18) and the resistance group (n=22). Both groups underwent two polysomnography tests, one at baseline and another after either a resistance training session (One Repetition Maximum - Strength Test, resistance group) or without physical exercise (control group).

DETAILED DESCRIPTION:
Upon completion of the baseline polysomnography (PSG), volunteers underwent body composition evaluations (total body mass, height and body mass index calculation) to characterize the sample. Three familiarization sessions were conducted with the exercise machines used in the study, and one repetition maximum test (1 RM) was completed in order to quantify the training session load. A PSG test was conducted on the same day of the exercise session for the resistance group, and the control group had a second PSG without exercise to compare the groups at both times.

The body composition assessment, the adaptations to the exercises and the training sessions were held at the Center for Psychobiology and Exercise Studies.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* sedentary lifestyle
* age between 65 and 80 years
* clinically good health (able to practice physical exercise)

Exclusion Criteria:

* known diseases of the cardiovascular, pulmonary, and musculoskeletal systems, diabetes
* profession in the field of physical exercise
* use of sleep medication
* disqualification based upon the clinical examination

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Sleep pattern measures in Polysomnography | The session of resistance training was performance about 16 hours before the polysomnographic

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Esteves, PhD, Principal Investigator — Universidade Federal de São Paulo; Valter AR Viana, MSc, Principal Investigator — Federal University of São Paulo; Marco Tulio de Mello, PhD, Study Chair — Federal University of São Paulo; Sergio Tufik, MD, PhD, Study Chair — Federal University of São Paulo; Rita A Boscolo, MSc, Principal Investigator — Federal University of São Paulo; Marcos G Santana, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Fderal de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Chasens ER, Sereika SM, Weaver TE, Umlauf MG. Daytime sleepiness, exercise, and physical function in older adults. J Sleep Res. 2007 Mar;16(1):60-5. doi: 10.1111/j.1365-2869.2007.00576.x. PMID 17309764
- [Result] Atkinson G, Davenne D. Relationships between sleep, physical activity and human health. Physiol Behav. 2007 Feb 28;90(2-3):229-35. doi: 10.1016/j.physbeh.2006.09.015. Epub 2006 Oct 25. PMID 17067643
- [Result] Cassilhas RC, Viana VA, Grassmann V, Santos RT, Santos RF, Tufik S, Mello MT. The impact of resistance exercise on the cognitive function of the elderly. Med Sci Sports Exerc. 2007 Aug;39(8):1401-7. doi: 10.1249/mss.0b013e318060111f. PMID 17762374